CLINICAL TRIAL: NCT05787457
Title: Comparative Metabolomics in Diabetes Patients From Sri Lanka and Switzerland
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-203/13; 2527 (Other: University Hospital Inselspital, Berne)
Record Dates: First submitted 2016-04-20; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Native South Asian population; Migrant South Asian population; Swiss ethnicity; Tamil ethnicity; Body fat distribution; Type 2 Diabetes; Magnetic resonance imaging; Genetic predisposition; Genetic background; Metabolomics; Non-targeted mass spectrometry; Insulin resistance; Hypertriglyceridaemia; Hyperinsulinaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Genetic Predisposition to Disease; Insulin Resistance; Hypertriglyceridemia; Hyperinsulinism | interventions — Restraint, Physical; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood (EDTA plasma, buffy coats and serum) samples are stored in Fluid X biobanking tubes. The tubes are labeled with a unique burnt-in 2D barcode and the respective plain digit number readable with magnifying glasses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tamil natives with Diabetes Type 2: Thirty Tamil natives (15 men, 15 women), representing general Tamil diabetic cohort.
  Interventions: Other: Clinical examination; Other: Blood testing; Other: MRI
- Swiss natives with Diabetes Type 2_matched: Thirty Swiss natives (15 men, 15 women) matching the Tamil cohort.
  Interventions: Other: Clinical examination; Other: Blood testing; Other: MRI
- Swiss natives with Diabetes Type 2_not matched: Thirty Swiss natives (15 men, 15 women), who are not matched to the Tamil cohort, representing general Swiss diabetic cohort.
  Interventions: Other: Clinical examination; Other: Blood testing; Other: MRI

INTERVENTIONS:
Other: Clinical examination
Other: Blood testing
Other: MRI

SUMMARY:
This study is a case-control study, where the assumed different subtypes of type 2 diabetes in people of Tamil ethnicity and Swiss origin living in Bern, Switzerland will be examined by measuring the metabolite profiles and the corresponding genetic background as well as ethnic differences in fat distribution performed by magnetic resonance imaging (MRI). The investigators aim to show that the specific metabolite profile and the fat distribution in the Tamil population is associated with the high prevalence of diabetes in this ethnicity. Fat distribution patterns are thought to determine the expression and severity of dysglycaemia. Additionally, the investigators aim to identify the key enzymes, their corresponding genes, and the respective polymorphisms relevant for these metabolic variations.

DETAILED DESCRIPTION:
Over the last two decades, the prevalence of type 2 diabetes has exploded among native and migrant South Asian populations. The earliest available epidemiological study in a rural sector in Sri Lanka showed a diabetes prevalence of 2.5% in 1990. In 2008 the Sri Lanka Diabetes, Cardiovascular Study (SLDCS) reported a prevalence of 10.3% for Sri Lankans aged ≥ 20 years. South Asian migrants living in western countries have higher diabetes prevalence rates compared with indigenous populations, around 10-14% in Europeans, 25-34% in Indian Asians. Moreover, type 2 diabetes develops at younger age in Asians than in Caucasian populations. In the UK the relative risk of type 2 diabetes in South Asian children is 14 times greater than in children of European descent.

A popular hypothesis for the greater prevalence of type 2 diabetes is that South Asians are undergoing rapidly changes in demographic profile, increasing urbanization and development and adoption of modern ("westernized") lifestyle. Nutrition transition, adoption of a sedentary lifestyle, reduced physical activity and possibly mental and social stress are held responsible for this increase. Especially the effect of dietary changes with higher intakes of sugars, animal fats and vegetable oils is large and most of the emerging epidemic of chronic disorders, like diabetes mellitus, are diet related. It has been detected that obesity induces excess lipolysis causing increased concentration of non-esterified fatty acids and triglycerides in blood and skeletal muscle. Lipotoxicity plays an important role in inducing insulin resistance and β-cell damage. Furthermore it has been observed that the kind of fat distribution correlates with the expression and the severity of dysglycaemia and that there are marked ethnic differences in fat distribution.

For example people of both South Asian and African Caribbean descent have an elevated risk of diabetes compared to Europeans. But while South Asians are centrally obese, dyslipidaemic and vulnerable to cardiac disease, African Caribbeans do not exhibit the diabetes related dyslipidaemic profile. A potential explanation for this discrepancy may lie in ethnic differences in fat distribution.

But it is not clear whether this can completely be attributed to ethnic differences, because features of insulin resistance, hypertriglyceridaemia, and hyperinsulinaemia are seen even in non-obese South Asian individuals. In contrast to Caucasian diabetic patients having a much higher BMI than the nondiabetic Caucasian population, the average BMI of Asians with diabetes is similar to the non-diseased population, indicating that South Asians diabetic patients in average are not obese. South Asians, however, have a much greater tendency to deposit intra-abdominal fat, which is metabolically active and strongly related to insulin resistance. Furthermore South Asians are proportionally fat due to less non-fat tissues. Therefore, insulin resistance in people of South Asian origin can occur even in the absence of conventionally defined obesity. The development of type 2 diabetes linked to obesity caused by overnutrition, which is regarded as a common feature in the Caucasian population, may not be typical in South Asians. This points at the limitations of BMI as a measure of adiposity across populations. These specific clinical characteristics, including a high degree of insulin resistance associated with abdominal fat deposition without massive obesity are common in patients of South Asian descent.

These findings suggest that Asians are more vulnerable than other ethnic groups to type 2 diabetes in response to a relatively small increase in body weight. Genetic susceptibility may be responsible for high prevalence of insulin resistance in South Asians . Such an escalating prevalence of type 2 diabetes is unlikely to be explained by genetic factors, indicating a greater influence of environmental factors in disease aetiology. Nevertheless type 2 diabetes has a strong genetic component. Most Asian diabetes patients have first-degree relative with diabetes. Several genetic variants have been identified by genome-wide association studies. Most genetic variants linked to type 2 diabetes seem to be related to insulin secretion rather than insulin resistance. In South Asian populations, however, the burden is the increased susceptibility to develop insulin resistance due to genetic predisposition and/or in response to certain environmental influences. These findings are showing the need for populations-specific studies. For this reason, the investigators restrict the study to the Tamil ethnic group living in Bern, Switzerland, with a Swiss reference cohort. The Tamil ethnicity is an isolated population with high prevalence of type 2 diabetes. Cultural customs have preserved this population from ethnic admixture. The first and the most of the second generation of migrated Tamils still belong to a population with a homogeneous genetic background, which facilitate to identify complex trait-susceptibility genes.

In contrast to many previous genome-wide association studies an inverse approach is taken for this study. The primary objective of this study is to show changes in the metabolic concentrations in plasma between Tamil individuals and native Swiss population using a mass-spectrometric approach. Type 2 diabetics have specific metabolic variations, and the investigators assume that South Asians and Caucasians differ in these alterations. The secondary aim of this study is to identify the key enzymes, their corresponding genes, and the respective polymorphisms relevant for the metabolic variations using a metabolic-pathway-based search including also intronic variants commonly missed by SNP (single nucleotide polymorphism)-and haplotype-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes per WHO criteria.
* Swiss ethnicity (defined as self-reported ancestry and parents and at least 1 grandparents are from Switzerland)
* Tamil ethnicity (defined as self-reported ancestry and parents and at least 1 grandparents are from Sri Lanka, belonging to ethnic identity of Tamils, respectively)
* Age limit: 18 - 75 years

Exclusion Criteria:

* Subjects with type 1 diabetes, steroid-induced diabetes, gestation diabetes, or pancreoprivic diabetes.
* Subjects with pregnancy.
* Subjects with metal implant, tattoos, or claustrophobia. MRI must be feasible.
* Subjects with severe chronic diseases, e.g. malignancies, heart or renal diseases (> stage 3).
* Subjects not able to provide informed consent.
* Enrolled in another study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of thirty Tamils and sixty native Swiss people with type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Metabolic phenotype of type 2 diabetes mellitus across groups | At baseline
  Significant metabolic changes in blood plasma of type 2 diabetic patients compared across groups as quantified by mass-spectrometric analysis

SECONDARY OUTCOMES:
Genetic Differences | At baseline
  Frequency of single nucleotide polymorphisms across groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fiedler, MD, MBA, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Sharing data depends on institutional (sponsor) and ethics agreement.

REFERENCES:
- [Background] Abate N, Carulli L, Cabo-Chan A Jr, Chandalia M, Snell PG, Grundy SM. Genetic polymorphism PC-1 K121Q and ethnic susceptibility to insulin resistance. J Clin Endocrinol Metab. 2003 Dec;88(12):5927-34. doi: 10.1210/jc.2003-030453. PMID 14671192
- [Background] Barnett AH, Dixon AN, Bellary S, Hanif MW, O'hare JP, Raymond NT, Kumar S. Type 2 diabetes and cardiovascular risk in the UK south Asian community. Diabetologia. 2006 Oct;49(10):2234-46. doi: 10.1007/s00125-006-0325-1. Epub 2006 Jul 18. PMID 16847701
- [Background] Ehtisham S, Crabtree N, Clark P, Shaw N, Barrett T. Ethnic differences in insulin resistance and body composition in United Kingdom adolescents. J Clin Endocrinol Metab. 2005 Jul;90(7):3963-9. doi: 10.1210/jc.2004-2001. Epub 2005 Apr 19. PMID 15840754
- [Background] Illangasekera U, Nugegoda DB, Perera LS. Prevalence of diabetes mellitus and impaired glucose tolerance in a rural Sri Lankan community. Ceylon Med J. 1993 Sep;38(3):123-6. PMID 7828231
- [Background] Illangasekera U, Rambodagalla S, Tennakoon S. Temporal trends in the prevalence of diabetes mellitus in a rural community in Sri Lanka. J R Soc Promot Health. 2004 Mar;124(2):92-4. doi: 10.1177/146642400412400214. PMID 15067982
- [Background] Jourdan C, Petersen AK, Gieger C, Doring A, Illig T, Wang-Sattler R, Meisinger C, Peters A, Adamski J, Prehn C, Suhre K, Altmaier E, Kastenmuller G, Romisch-Margl W, Theis FJ, Krumsiek J, Wichmann HE, Linseisen J. Body fat free mass is associated with the serum metabolite profile in a population-based study. PLoS One. 2012;7(6):e40009. doi: 10.1371/journal.pone.0040009. Epub 2012 Jun 27. PMID 22761945
- [Background] Katulanda P, Constantine GR, Mahesh JG, Sheriff R, Seneviratne RD, Wijeratne S, Wijesuriya M, McCarthy MI, Adler AI, Matthews DR. Prevalence and projections of diabetes and pre-diabetes in adults in Sri Lanka--Sri Lanka Diabetes, Cardiovascular Study (SLDCS). Diabet Med. 2008 Sep;25(9):1062-9. doi: 10.1111/j.1464-5491.2008.02523.x. PMID 19183311
- [Background] Katulanda P, Sheriff MH, Matthews DR. The diabetes epidemic in Sri Lanka - a growing problem. Ceylon Med J. 2006 Mar;51(1):26-8. doi: 10.4038/cmj.v51i1.1373. PMID 16898034
- [Background] Ramachandran A, Ma RC, Snehalatha C. Diabetes in Asia. Lancet. 2010 Jan 30;375(9712):408-18. doi: 10.1016/S0140-6736(09)60937-5. Epub 2009 Oct 28. PMID 19875164
- [Background] Unger RH, Zhou YT. Lipotoxicity of beta-cells in obesity and in other causes of fatty acid spillover. Diabetes. 2001 Feb;50 Suppl 1:S118-21. doi: 10.2337/diabetes.50.2007.s118. PMID 11272168
- [Background] Vandenheede H, Deboosere P, Stirbu I, Agyemang CO, Harding S, Juel K, Rafnsson SB, Regidor E, Rey G, Rosato M, Mackenbach JP, Kunst AE. Migrant mortality from diabetes mellitus across Europe: the importance of socio-economic change. Eur J Epidemiol. 2012 Feb;27(2):109-17. doi: 10.1007/s10654-011-9638-6. Epub 2011 Dec 14. PMID 22167294